CLINICAL TRIAL: NCT03675984
Title: Development of Exercise Protocol for Scoliosis Using Surface Electromyography(S-EMG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ju Seok Ryu (Other)
Responsible Party: Sponsor-Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1701/378-103
Record Dates: First submitted 2018-09-10; First posted 2018-09-18 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Scoliosis
Keywords: surface EMG, cobb angle, exercise, Spinal Curvatures
MeSH Terms: conditions — Motor Activity; Spinal Curvatures

STUDY DESIGN:
Intervention Model Description: Annual evaluation after educating asymmetrical stabilization exercise. Cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- asymmetrical stabilization exercise group (Experimental): 'asymmetrical stabilization exercise' patient learn asymmetrical stabilization exercise according to the asymmetrical paraspinal muscles weakness and curve type
  Interventions: Behavioral: asymmetrical stabilization exercise

INTERVENTIONS:
Behavioral: asymmetrical stabilization exercise — Exercise is combined to form an appropriate combination of motion (Side-lying, Bird-dog, Prone arm lift, Prone leg lift) according to the curve pattern and muscle weakness of each patient's.

SUMMARY:
There has been much effort in recent years to better understand the causes of idiopathic scoliosis (IS). Some studies suggested muscle imbalance as a cause of scoliosis based on asymmetric muscular activation. Surface electromyography can evaluate asymmetrical muscular weakness. Therefore, the peak amplitude values can be used to compare the side to side differences in paraspinal muscles. From these findings the investigators improve the exercise method of IS according to muscle weakness and curve pattern.

DETAILED DESCRIPTION:
Design: Prospective study Setting: hospital rehabilitation department the investigators will check the muscular activation at bilateral paraspinal muscles with surface electromyography and curve type with simple radiography.

Intervention: After that the investigators educate asymmetrical stabilization exercise according to muscle weakness and curve pattern.

Main outcome measures: Cobb angle

ELIGIBILITY:
Inclusion Criteria:

* X-ray shows a cobb angle of 10 degrees or higher.
* Patients 8 and older.

Exclusion Criteria:

* Patients with spinal surgery
* Patients with scoliosis caused by cerebral palsy, muscle paralysis, polio, congenital spinal cord abnormalities, etc.
* Cobb angle less than 10 degrees and more than 40 degrees
* Patients with acute back pain

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Cobb angle | through study completion, an average of 6 months
  the angle of curvature be measured by drawing lines parallel to the upper border of the upper vertebral body and the lower border of the lowest vertebra of the structural curve on plain radiography

SECONDARY OUTCOMES:
Scoliosis Research Society-22(SRS-22) | through study completion, an average of 6 months
  questionnaire for evaluating quality of life in patients with idiopathic scoliosis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyungji-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes